CLINICAL TRIAL: NCT05036772
Title: Assessment of Patients' Pain and Anxiety During a Hysterosalpingography Narratified by a Virtual Reality Helmet.
Brief Title: Assessment of Patients' Pain and Anxiety During a Hysterosalpingography Narratified by a Virtual Reality Helmet (Daphné)
Acronym: Daphné
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Daphné
Record Dates: First submitted 2021-07-05; First posted 2021-09-08 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-03

CONDITIONS: Salpingography; Virtual Reality Exposure Therapy; Virtual Reality; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Practice (No Intervention): The control arm is supported according to the usual practice. The experimental arm will have the possibility to use a distracting virutel environment for the duration of hysterosalpingography
- Interventionnal (Experimental): The experimental arm will have the possibility to use a distracting virutel environment for the duration of hysterosalpingography.
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — The experimental arm will have the possibility to use a distracting virutel environment for the duration of hysterosalpingography.
  Arms: Interventionnal

SUMMARY:
Compare the maximum pain and anxiety experienced between the group using a virtual reality headset and the control group in an adult woman during a hysterosalpingography examination

DETAILED DESCRIPTION:
In France, 1 couples out of 5 consults for suspected infertility. Hysterosalpingography is the first line diagnostic examination in this course and can sometimes be therapeutic. This gynecological examination is invasive in nature, this exam requires an administration of iodinated contrast product by the endocavitary route.

Hysterosalpingography is the most painful examination in this treatment path and pain's assessment is classified as strong by the French National Authority for Health (Haute Autérité de Santé) and anxiety-inducing. For these patients, drug analgesic treatments remain ineffective or contraindicated in outpatient mode. Ionizing irradiation is a constraint that makes hypnosis unsuitable.

Several studies show the contribution of a virtual reality headset in reducing pain and anxiety by inducing patients in an hypnotic environment. This tool standardizes interventions based on changes in consciousness. It is an easy-to-use, non-drug analgesia with few side effects and inexpensive.

The environment offered by this medical device is based on evidence to peacefully escort patients on a journey of natural elements. Calm music is made up of key elements of musical therapy. A medical anesthesiologist and hypnotherapist wrote the hypnotic induction. And, the voice is the one of an experienced sociologist in practice. A simple meditation modeled on heart synchronization sets a persistent goal during this immersion.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* patients with a prescription for hysterosalpingography
* patients able to answer the questionnaire independently (French-speaking or understanding French)
* informed consent, signed by the patient
* patients benefiting from a social security scheme or benefiting through a third party

Exclusion Criteria:

* patients with a contraindication to virtual reality headset.
* refusal to participate in the study
* Contraindication to the realization of hysterosalpingography (pregnancy / lactation or infection)
* patient under guardianship, curatorship or subordination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
visual analog scale (EVA) | through study completion, an average of 1 year
  The patient rates her pain level between 0 and 10. The standard question is: "From 0 to 10, with 0 absence of pain and 10 maximum pain, how much will you rate the maximum pain experienced during your examination?"

SECONDARY OUTCOMES:
anxiety assessment | through study completion, an average of 1 year
  State Trait Inventory Anxiety (STAI Y-A) anxiety assessment questionnaire
Dosimetry | through study completion, an average of 1 year
  Collection of the dose report produced surface in mGy.cm²
Time of exam | through study completion, an average of 1 year
  Measurement of the time in minutes between the first shot and the last shot (the late evacuation shot will not be taken into account)
- Cybersickness evaluation | through study completion, an average of 1 year
  simplified Virtual Reality Sickness Questionnaire (VRSQ) cybersickness scale. (Questionnaire in 9 items)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Poitiers, France

IPD SHARING:
Plan to Share IPD: No